CLINICAL TRIAL: NCT01171599
Title: PACE-CALL: A Weight Control Intervention for Survivors of Childhood Leukemia
Acronym: PACE-CALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Kevin Patrick, MD, MS, University of California, San Diego
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R21CA128019 (NIH)
Record Dates: First submitted 2010-07-23; First posted 2010-07-28 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Overweight; Weight Loss; Weight Maintenance
Keywords: Weight Loss; Obesity; Overweight; Physical Activity; Nutrition; Youth; Adolescent; Technology
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Fit4Life — As previously described, the purpose of this study is to develop a web and text message based weight loss intervention for childhood acute lymphoblastic leukemia survivors (ALL) survivor. The web and text message based intervention that is being developed will be evaluated in a separate ACS (American Cancer Society) funded trial randomized control trial. The web and text message based intervention (there are other intervention features that do not relate to the web & text based platforms that were developed as part of this NIH funded study) is a 16-week program that includes:

SUMMARY:
The purpose of this National Cancer Institute (NCI) funded study is to develop and test the acceptability and usability of a web & text message based weight loss intervention for childhood acute lymphoblastic leukemia (ALL) survivors. Childhood cancer survivors ages 7 - 18 will provide feedback during focus groups on a web and text message based program that was developed.

DETAILED DESCRIPTION:
This is a two year study to develop a predominantly web-based behavioral assessment and intervention program (PACE-CALL) that will provide individual assessment and tailoring of a behavioral intervention for adolescent children Acute Lymphoblastic Leukemia (ALL) survivors and their families. In addition, we are conducting formative research to adapt the abovementioned program to children and adolescents aged 7 - 18 who survived any cancer.

Focus Groups: Web-Based & Text Message Intervention Feedback

Two focus groups will be conducted with adolescent cancer survivors and their families, to assess the usability and acceptability of the web-based intervention, focus groups will be conducted. The two focus groups will last 2 hours with 6-8 people in each group: one focus group with youth & adolescents (age 7 - 18 who are representative of the target population to determine the appropriateness of the web-based intervention one focus group with the parents of the children in the focus group mentioned above (it will occur at the same time). All focus groups will begin with an overview of the study and description of the web-based intervention components. Focus group participants will see sample web pages and may be asked to provide feedback on some or all of the following:

Youth, Adolescent or Parent:

* How does the web-based and text message based intervention address issues faced by children who have survived cancer?
* What do you like about the web-based intervention? What do you not like about the web-based intervention? What would you change about the web-based intervention?
* What do you like about the text messages? What do you not like about the text messages?
* Would you want to join a program like this? Why or why not?
* If you were to be in this program, how often would you log on to the web-based intervention? How often would you want to receive text messages?
* What are some of the barriers to joining a program like this?

ELIGIBILITY:
Inclusion Criteria:

* Are 7 - 18 years
* Provide assent and have a legal guardian that will participate and provide parental permission/consent
* Are a cancer survivor (off treatment for two years)
* Are overweight or obese (85th percentile BMI (Body Mass Index) for age and gender)

Exclusion Criteria:

* Have any of the following comorbidities of obesity that require immediate sub-specialist referral including pseudotumor cerebri, sleep apnea, and obesity hypoventilation syndrome

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Acceptability and Usability of a Web & Text Message Based Intervention through Qualitative Feedback from Focus Groups | 2-hour focus group
  The primary outcome is to develop a web and text message based weight loss intervention that will provide individual assessment and tailoring of a behavioral intervention for ALL survivors. In order to test the acceptaibility and usability of the website and text message program, focus groups will be conducted with cancer survivors to provide feedback on the program.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD
Locations (1):
- UCSD, Atkinson Hall, 3rd Floor, La Jolla, California, United States